CLINICAL TRIAL: NCT04146467
Title: A Prospective, Multi-Center, Evaluator-Blinded Study Evaluating the Safety and Effectiveness of the Renuvion APR Device to Improve the Appearance of Lax Tissue in the Neck and Submental Region
Brief Title: Renuvion APR Device to Improve the Appearance of Lax Tissue in the Neck and Submental Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VP-1902
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Lax Skin
Keywords: Submental, Neck
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Study Phase I (Experimental): Subjects will be treated with the Renuvion APR device in the neck and submental region.
  Interventions: Device: Renuvion APR Device
- Study Phase II (Experimental): Subjects will be treated with the Renuvion APR device in the neck and submental region.
  Interventions: Device: Renuvion APR Device

INTERVENTIONS:
Device: Renuvion APR Device — The Renuvion APR Handpiece is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with compatible generators for the percutaneous delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue. Radiofrequency energy is delivered to the handpiece by the generator and used to energize the electrode. When helium gas is passed over the energized electrode, a helium plasma is generated for soft tissue cutting, coagulation or ablation. The Renuvion APR Handpiece has a non-extendable electrode to generate helium plasma.

SUMMARY:
This is a prospective, multi-center, multi-phase, evaluator-blinded study of subjects undergoing a procedure with the Renuvion APR Device to improve the appearance of lax tissue in the neck and submental region.

DETAILED DESCRIPTION:
This is a prospective, multi-center, multi-phase, evaluator-blinded study of subjects undergoing a procedure to improve the appearance of lax tissue in the neck and submental region. All study subjects will be treated with the Renuvion APR Device.

Phase I (n=17) of this study will be conducted primarily to provide safety data, however, effectiveness data will also be collected at the above stated timepoints through 6 months post-procedure.

Phase II (n=65) of this study is the expansion of the study to a pivotal study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 35-65 years of age (inclusive).
2. Healthy as determined by the investigator examining the subject.
3. Seeking improvement of the appearance of lax tissue in the neck and submental region.
4. Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation.
5. Willing and able to comply with protocol requirements, including obtaining study-required images/photos and assessments, and returning for follow-up visits.
6. Willing to release rights for the use of study photos, including in potential publication.
7. Understands and accepts the obligation not to have significant weight loss or weight gain (≥8 pounds) post the treatment, and for the duration of participation in the study.
8. Willing to abstain from the use of blood thinners (including, but not limited to, Coumadin, NSAIDS, Ibuprofen, vitamin K, other) for 2 weeks (14 days) prior to the procedure.
9. Willing to abstain from smoking, vaping, or the use of e-cigarettes for 1 year prior to and for the entire duration of participation in the study.
10. Willing to abstain from the use of marijuana for 2 weeks prior to and for the duration of participation in the study.
11. Able to read, understand, sign and date the informed consent document (English only).

Exclusion Criteria:

1. Pregnant or lactating.
2. Pregnancy within 12 months prior to screening.
3. Use within 24 hours preceding surgery of ibuprofen, acetaminophen, any other analgesics, anti-inflammatory products, or any products including herbals and supplements that could interfere with the clinical assessments of this study (other than drugs used for anesthesia).
4. Allergy to tumescent anesthetic (lidocaine/epinephrine).
5. Excessive subcutaneous fat in the treatment area (as determined by the treating investigator).
6. Active systemic or local skin disease that may alter wound healing.
7. Significant or uncontrolled medical condition that, in the opinion of the investigator, participation in the study may compromise the patient's health.
8. Severe solar elastosis.
9. History of autoimmune disease (excluding Hashimoto's thyroiditis).
10. Known hypersensitivity or adverse reaction to anesthetics.
11. Known susceptibility to keloid formation or hypertrophic scarring.
12. Cancerous or pre-cancerous lesions in the area to be treated.
13. History or current diagnosis of cancer of any type (excluding skin cancer).
14. History of uncontrolled cardiovascular disease (i.e. myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other).
15. History, or current bleeding disorders (i.e. hemophilia or von Willebrand disease), or anticipated treatment with prescription anticoagulants.
16. Possesses a surgically implanted electronic device (i.e. pacemaker).
17. History of AIDs/HIV.
18. Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
19. Chronic hypoxia or dependence on supplemental oxygen.
20. Participation in any other investigational study within 30 days prior to consent.
21. Any surgical or transdermal neck/submental aesthetic procedures or plans to undergo any other aesthetic procedure during study participation. Such procedures include, but are not limited to, submentoplasty, liposuction, ultrasound, cryolipolysis, radiofrequency, and laser.
22. History of or current injury to the head and neck or any area of the body being treated as a part of this study.
23. Presence of more than mild platysmal banding as per the Geister, et al Validated Assessment Scale for Platysmal Bands.
24. Subject requiring removal of adipose tissue prior index procedure.
25. A family member of the investigator or sponsor; an employee of the investigator or sponsor.
26. Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Ruff IV, MD, Principal Investigator — West End Plastic Surgery
Locations (6):
- United States (6):
  - Faces+ Plastic Surgery, San Diego, California
  - West End Plastic Surgery, Washington D.C., District of Columbia
  - New Jersey Clinical Research Center, Montclair, New Jersey
  - Luxurgery, New York, New York
  - H/K/B Cosmetic Surgery, Huntersville, North Carolina
  - Facial Plastic & Aesthetic Laser Center, Youngstown, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Sub-Dermal Neck Renuvion APR Device - Study Phase I; Sub-Dermal Neck Renuvion APR Device - Study Phase II: All subjects will be treated with the Renuvion APR device.
  Renuvion APR Device: The Renuvion APR Handpiece is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with compatible generators for the percutaneous delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue. Radiofrequency energy is delivered to the handpiece by the generator and used to energize the electrode. When helium gas is passed over the energized electrode, a helium plasma is generated for soft tissue cutting, coagulation or ablation. The Renuvion APR Handpiece has a non-extendable electrode to generate helium plasma.
Period: Overall Study
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Started | 17 | 65
Completed | 17 | 62
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II | Total
Number analyzed (Participants) | 17 | 65 | 82
Age, Customized [Mean (Standard Deviation); unit: years]
  Average Age | 58.5 (4.0) | 55.9 (6.3) | 56.4 (5.9)
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Median Age | 59 [56 to 62] | 57.0 [51 to 61] | 57.0 [53 to 61.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 59 | 75
  Male | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Hispanic or Latino | 1 | 3 | 4
  White | 14 | 61 | 75
  Other: Greek Spanish | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 17 | 65 | 82
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 36.49 (4.1) | 25.4 (4.9) | 25.5 (4.7)
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 25.5 [22.6 to 28.3] | 24.7 [22.8 to 27.0] | 24.8 [22.7 to 27.6]

OUTCOME MEASURES:

1. Primary Outcome: Day 180 Number of Participants With Improvement Measured By Independent Photographic Review
Description: Improvement in the appearance of lax tissue in the neck and submental region at 6 months as determined by qualitative 2D photography assessment by blinded Independent Photographic Reviewers. Three experienced, blinded photographic reviewers performed a qualitative analysis/review of the pre-treatment and post-treatment sets of images of each subject in a blinded and randomized order. Each blinded reviewer chose which image was the post-treatment image. Success was correct post-treatment image selection by at least 2 of the 3 reviewers. The percentage of subjects with a correct post-treatment image selection was calculated.
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Groups:
- Sub-Dermal Neck Renuvion APR Device - Study Phase II: All subjects treated with the Renuvion APR device.
  Renuvion APR Device: The Renuvion APR Handpiece is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with compatible generators for the percutaneous delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue. Radiofrequency energy is delivered to the handpiece by the generator and used to energize the electrode. When helium gas is passed over the energized electrode, a helium plasma is generated for soft tissue cutting, coagulation or ablation. The Renuvion APR Handpiece has a non-extendable electrode to generate helium plasma.
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 7 | 63
Participants | 6 | 52
Statistical Analysis 1: Comparison: Sub-Dermal Neck Renuvion APR Device - Study Phase II; Test type: Superiority; p < 0.0001, Fisher Exact

2. Primary Outcome: Subject Reported Pain - None to Moderate
Description: The primary safety endpoint is the level of pain and discomfort after treatment as reported by the subject on an 11-point Numeric Rating Scale (NRS) through the 7-day follow-up visit where 0 is no pain and 10 is the most pain. Pain scores are classified as scores of 0 being no pain, 1 - 5 is minor pain, 6 - 7 is moderate pain, and 8 - 10 is severe pain.
  The primary safety objective is to demonstrate that the proportion of subjects with none-to- moderate pain exceeds the performance goal (PG). The performance goal is 55%.
Time Frame: Day 7
Population: Phase I: 17 total participants started Phase I. 4 participants missed their Day 7 follow-up visit due to COVID-19 office closures and/or restrictions. Therefore, Day 7 data for Subject Reported Pain was only analyzed for 13 participants.
  Phase II: 65 participants started Phase 2. 1 participant exited the study prior to Day 7 follow-up visit. Therefore, Day 7 data for Subject Reported Pain was only analyzed for 64 participants.
Measure: Count of Participants; unit: Participants
Groups:
- Sub-Dermal Neck Renuvion APR Device - Study Phase I: All subjects treated with the Renuvion APR device.
  Renuvion APR Device: The Renuvion APR Handpiece is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with compatible generators for the percutaneous delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue. Radiofrequency energy is delivered to the handpiece by the generator and used to energize the electrode. When helium gas is passed over the energized electrode, a helium plasma is generated for soft tissue cutting, coagulation or ablation. The Renuvion APR Handpiece has a non-extendable electrode to generate helium plasma.
- Sub-Dermal Neck Renuvion APR Device - Study Phase II: Subjects treated with the Renuvion APR device.
  Renuvion APR Device: The Renuvion APR Handpiece is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with compatible generators for the percutaneous delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue. Radiofrequency energy is delivered to the handpiece by the generator and used to energize the electrode. When helium gas is passed over the energized electrode, a helium plasma is generated for soft tissue cutting, coagulation or ablation. The Renuvion APR Handpiece has a non-extendable electrode to generate helium plasma.
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 13 | 64
Participants | 13 | 62

3. Other Pre Specified Outcome: Day 90 Number of Participants With Improvement Measured By Independent Photographic Review
Description: Change in the appearance of lax tissue in the neck and submental region at 90-days as determined by qualitative 2D photography assessment by blinded Independent Photographic Reviewers. Three experienced, blinded photographic reviewers performed a qualitative analysis/review of the pre-treatment and post-treatment sets of images of each subject in a blinded and randomized order. Each blinded reviewer chose which image was the post-treatment image. Success was correct post-treatment image selection by at least 2 of the 3 reviewers. The percentage of subjects with a correct post-treatment image selection was calculated.
Time Frame: 90-Day
Population: Phase I: 17 total participants started Phase I. 7 participants missed their D90 images due to COVID-19 office closures and/or restrictions. Therefore, D90 Independent Photographic Review data was only available for 10 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D90 visit and 1 participant was lost to follow-up prior to D90 Follow-up visit. Therefore, Day 90 Independent Photographic Review data was only available for 63 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 10 | 63
Participants | 8 | 48
Statistical Analysis 1: Comparison: Sub-Dermal Neck Renuvion APR Device - Study Phase II; Test type: Superiority; p < 0.0004, Fisher Exact

4. Other Pre Specified Outcome: Subject Modified Global Aesthetic Improvement Scale (GAIS)
Description: Subject Modified GAIS: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: 90-Day
Population: Phase I: 17 total participants started Phase I. 1 participant missed their D90 Modified GAIS due to COVID-19 office closures and/or restrictions. Therefore, D90 Subject Modified GAIS data was only available for 16 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D90 visit and 1 participant was lost to follow-up prior to D90 Follow-up visit. Therefore, Day 90 Subject Modified GAIS data was only available for 63 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 16 | 63
Participants
  Very Much Improved | 0 | 7
  Much Improved | 7 | 18
  Improved | 5 | 33
  No Change | 3 | 3
  Worse | 0 | 1
  Much Worse | 0 | 1
  Very Much Worse | 1 | 0

5. Other Pre Specified Outcome: Subject Modified Global Aesthetic Improvement Scale (GAIS)
Description: Subject Modified GAIS: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: 180-Day
Population: Phase-II discrepancy is due to 1 subject exited due to an AE during treatment and 2 subject lost to follow-up prior to Day 180 visit. Which brought the numbers to: Phase-II 62
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 17 | 62
Participants
  Very Much Improved | 4 | 12
  Much Improved | 5 | 17
  Improved | 3 | 24
  No Change | 3 | 7
  Worse | 1 | 2
  Much Worse | 0 | 0
  Very Much Worse | 1 | 0

6. Other Pre Specified Outcome: Investigator Modified Global Aesthetics Improvement Scale (GAIS)
Description: Investigator Modified GAIS:Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: 90-Day
Population: Phase I: 17 total participants started Phase I. 2 participants completed virtual visits and 1 participant missed their D90 visit due to COVID-19 office closures and/or restrictions. Therefore, D90 Investigator GAIS data was only available for 14 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D90 visit and 1 participant was lost to follow-up prior to D90 visit. Therefore, Day 90 Investigator GAIS data was only available for 63 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 14 | 63
Participants
  Very Much Improved | 0 | 8
  Much Improved | 3 | 19
  Improved | 8 | 33
  No Change | 2 | 3
  Worse | 1 | 0
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

7. Other Pre Specified Outcome: Investigator Modified Global Aesthetic Improvement Scale (GAIS)
Description: Investigator Modified GAIS: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: 180-Day
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 17 | 62
Participants
  Very Much Improved | 2 | 8
  Much Improved | 6 | 19
  Improved | 5 | 27
  No Change | 3 | 6
  Worse | 1 | 2
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

8. Other Pre Specified Outcome: Day 180 Patient Satisfaction Questionnaire (PSQ) of Procedure
Description: At 180 days post procedure, the subject's satisfaction with the procedure was assessed using a Patient Satisfaction Questionnaire. Questions were YES or NO questions pertaining to satisfaction with study treatment, observations of improvement, and considerations for recommendation.
Time Frame: 180-Day
Population: Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D180 visit and 2 participants was lost to follow-up prior to D180 Follow-up visit. Therefore, Day 180 Patient Satisfaction Questionnaire data was only available for 62 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 17 | 62
Participants
  Number of Subjects that Answered YES to Happy With Results of Procedure | 12 | 47
  Number of Subjects that Answered YES to More Jawline Definition | NA — Data not collected in Study Phase I | 39
  Number of Subjects that Answered YES to Reduction in Jowls | NA — Data not collected in Study Phase I | 20
  Number of Subjects that Answered YES to Improvement in Skin Texture in Treatment Area | NA — Data not collected in Study Phase I | 20
  Number of Subjects that Answered YES to Reduction in the Area Under the Chin | NA — Data not collected in Study Phase I | 41
  Number of Subjects that Answered YES to Reduction of Lines & Wrinkles in the Treatment Area | NA — Data not collected in Study Phase I | 21
  Number of Subjects that Answered YES to Other Changes | NA — Data not collected in Study Phase I | 10
  Number of Subjects that Answered YES to Would Recommend Procedure to a Friend | 12 | 46
  Number of Subjects that Answered YES to Would Consider Having the Procedure on Another Body Area | 11 | 47

9. Other Pre Specified Outcome: Quantitative Improvement in Overall Lift of the Neck and Submental Area
Description: Quantitative improvement in overall lift of the neck and submental area as determine by quantitative assessment based on 2D photography with Canfield Vectra system analysis. Fixed landmarks on the subject's face were used.
Time Frame: 180-Day
Population: Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D180 visit, 1 participant completed a virtual visit, and 2 participants were lost to follow-up prior to D180 Follow-up visit. Therefore, Day 180 Quantitative Improvement data was only available for 61 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 0 | 61
Participants |  | 38

10. Other Pre Specified Outcome: Quantitative Improvement in Submental Volume
Description: Quantitative improvement in submental volume at 180 days as determined by quantitative assessment based on 3D photography with Canfield Vectra system analysis.
Time Frame: 180-Day
Population: Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D180 visit, 2 participants were lost to follow-up prior to D180 visit, 1 participant completed a virtual visit for D180 and did not have photographs for volume assessment, and 1 subject had poor image quality that resulted in the inability to assess volume change. Therefore, Day 180 Quantitative Improvement in Submental Volume was only available for 60 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 0 | 60
Participants |  | 41

11. Other Pre Specified Outcome: Average Pain at Day 7 Reported by Subject
Description: Level of pain and discomfort after treatment as reported by the subject on a 11-point Numeric Rating Scale where 0 is "No Pain" and 10 is "Worst Possible Pain"
Time Frame: 7-Day
Population: Phase I: 17 total participants started Phase I. 4 participants missed their D7 follow-up visit due to COVID-19 office closures and/or restrictions. Therefore, D7 Average Pain data was only available for 13 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D7 visit . Therefore, Day 7 Average Pain data was only available for 64 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 13 | 64
score on a scale | 1.23 (1.24) | 0.6 (1.2)
Statistical Analysis 1: Comparison: Sub-Dermal Neck Renuvion APR Device - Study Phase II; Test type: Superiority; p < 0.0001, Fisher Exact

12. Other Pre Specified Outcome: Median Pain Reported by Subject at Day 7
Description: as for outcome 11
Time Frame: 7-Day
Population: Phase I: 17 total participants started Phase I. 4 participants missed their D7 follow-up visit due to COVID-19 office closures and/or restrictions. Therefore, D7 Median Pain data was only available for 13 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D7 visit . Therefore, Day 7 Median Pain data was only available for 64 participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 13 | 64
score on a scale | 1.0 [0 to 3] | 0.0 [0 to 1]

13. Other Pre Specified Outcome: Average Pain Reported by Subject at Day 30
Description: as for outcome 11
Time Frame: 30-Day
Population: Phase I: 17 total participants started Phase I. 2 participants missed their D30 follow-up visit due to COVID-19 office closures and/or restrictions. Therefore, D30 Average Pain data was only available for 15 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D30 visit and1 participant was lost to follow-up prior to D30 visit. Therefore, Day 30 Average Pain data was only available for 63 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 15 | 63
score on a scale | 1.33 (2.66) | 0.2 (0.5)

14. Other Pre Specified Outcome: Median Pain Reported by Subject at Day 30
Description: as for outcome 11
Time Frame: 30-Day
Population: Phase I: 17 total participants started Phase I. 2 participants missed their D30 follow-up visit due to COVID-19 office closures and/or restrictions. Therefore, D30 Median Pain data was only available for 15 participants.
  Phase II: 65 total participants started Phase 2. 1 participant exited the study prior to D30 visit and1 participant was lost to follow-up prior to D30 visit. Therefore, Day 30 Median Pain data was only available for 63 participants.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase I | Sub-Dermal Neck Renuvion APR Device - Study Phase II
Number analyzed (Participants) | 15 | 63
score on a scale | 0 [0 to 9] | 0.0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Through 6 month follow-up visit for all enrolled subjects
Arm/Group | Sub-Dermal Neck Renuvion APR Device - Study Phase II | Sub-Dermal Neck Renuvion APR Device - Study Phase I
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/17
Serious Adverse Events (participants affected / at risk) | 3/65 | 0/17
Other Adverse Events (participants affected / at risk) | 62/65 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub-Dermal Neck Renuvion APR Device - Study Phase II (N=65) | Sub-Dermal Neck Renuvion APR Device - Study Phase I (N=17)
Lower GI Bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not related to device or procedure.
Acute Appendicitis (General disorders) | 1 (1) | 0 (0) — Not related to device or procedure.
Kidney Stone (Renal and urinary disorders) | 1 (1) | 0 (0) — Not related to device or procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sub-Dermal Neck Renuvion APR Device - Study Phase II (N=65) | Sub-Dermal Neck Renuvion APR Device - Study Phase I (N=17)
Edema/Swelling (Skin and subcutaneous tissue disorders) | 60 | 14 — Expected Treatment Effect
Temporary sensory nerve injury (loss of sensation) (Skin and subcutaneous tissue disorders) | 57 | 5 — Expected Treatment Effect
Ecchymosis/ bruising (Skin and subcutaneous tissue disorders) | 36 | 10 — Expected Treatment Effect
Erythema (Skin and subcutaneous tissue disorders) | 32 | 3 — Expected Treatment Effect
Crepitus (Skin and subcutaneous tissue disorders) | 27 | 3 — Expected Treatment Effect
Pain/tenderness (Skin and subcutaneous tissue disorders) | 16 | 5 — Expected Treatment Effect
Nodules/subcutaneous lumps (migratory firmness) (Skin and subcutaneous tissue disorders) | 8 | 6 — Expected Treatment Effect
Temporary motor nerve Injury (nerve weakness, muscle atrophy, twitching, and paralysis) (Nervous system disorders) | 4 | 1
Pruritus/itching (not related to nerve injury) (Skin and subcutaneous tissue disorders) | 4 | 0

LIMITATIONS AND CAVEATS:
Limitations of this study was the pandemic that occurred in the middle of the study and caused study visits to be more challenging for all subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04146467/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT04146467/SAP_001.pdf